CLINICAL TRIAL: NCT03327311
Title: Histological Analysis of Bellafill Injected Tissue at Various Time Points: A Proof of Concept Study
Brief Title: Histological Analysis of Bellafill Injected Tissue at Various Time Points
Status: Completed | Type: Observational
Sponsor: Suneva Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SUN-1502
Record Dates: First submitted 2015-12-29; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Histopathology
Keywords: No condition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue Pathology
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Bellafill 1 week post-injection: n=2. Histopathology conducted 1 week post-injection
  Interventions: Device: Bellafill
- Bellafill 1 month post-injection: n=2. Histopathology conducted 1 month post-injection
  Interventions: Device: Bellafill
- Bellafill 2 months post-injection: n=2. Histopathology conducted 2 months post-injection
  Interventions: Device: Bellafill
- Bellafill 3 months post-injection: n=2. Histopathology conducted 3 months post-injection
  Interventions: Device: Bellafill
- Bellafill 6 months post-injection: n=2. Histopathology conducted 6 months post-injection
  Interventions: Device: Bellafill

INTERVENTIONS:
Device: Bellafill — Bellafill injected into site of pre-planned surgery (i.e., mini-abdominoplasty or redundant abdominal tissue removal) at two depths (dermis & deep dermis).

SUMMARY:
This is a prospective, in vivo proof-of-concept clinical study, where histopathologic examinations will be conducted at various timepoints following Bellafill injections.

DETAILED DESCRIPTION:
Visit 1 (day 0): Subjects with pre-planned surgical treatment (mini-abdominoplasty or redundant abdominal tissue removal) will be enrolled and will receive a Bellafill Skin Test.

Visit 2 (Day 28): Each subject receives treatment with Bellafill into 2 identified rectangular treatment areas within the pre-planned surgical area (0.1cc injected in the upper dermis and 0.1cc injected in the deep dermis at the subcutaneous junction).

Visit 3 (1 Week, 1 Month, or 2 Months; or, 3 Months or 6 Months): The timing of Visit 3 (the final study visit) is dependent on the subject's type of pre-planned surgery. Subjects who will undergo abdominoplasty will attend Visit 3 at 1 Week, 1 Month or 2 Months after Visit 2. Subjects who will undergo removal of redundant skin (i.e., dog ear) will attend Visit 3 at 3 Months or 6 Months after Visit 2. Following surgical removal of Bellafill injection sites, histopathologic analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Female or male in good general health greater than 21 years of age. Female Subjects of childbearing potential must have a negative urine pregnancy test result at Baseline and practice a reliable method of contraception throughout the study.
* Subject must sign an IRB-approved Informed Consent Form, Photographic Release Form, California Experimental Subject's Bill of Rights Form and the Authorization for Use and release of Health and Research Study Information (HIPAA) form prior to any study-related procedures being performed.
* Fitzpatrick skin type I-III.
* Planned adominoplasty surgery or post tummy- tuck surgery for redundant skin ("dog ear") removal surgery.
* Sufficient adominoplasty tissue or redundant skin ("dog ear") to allow for planned tissue procurement.
* Willing to comply with study protocols and complete the entire course of the study.

Exclusion Criteria:

* A female subject that is pregnant (positive UPT), breast-feeding, or who is of childbearing potential and not practicing a reliable method of birth control.
* Positive Bellafill Skin Test
* Any skin pathology or condition that could interfere with the evaluation of the treatment areas, worsen due to the proposed treatment or require interfering topical, systemic or surgical therapy.
* Have a recent or current history of inflammatory skin disease, infection, cancerous/pre-cancerous lesion, unhealed wound or clinically significant acne in the proposed biopsy areas.
* History of systemic granulomatous diseases active or inactive (e.g., Sarcoid, Wegeners, TB, etc.) or connective tissue diseases (e.g., lupus, dermatomyositis, etc.).
* History of any previous injectable filler to the study treatment area.
* Have known susceptibility to keloid formation or hypertrophic scarring.
* History of Bleeding Disorders.
* Known hypersensitivity or previous allergic reaction to any of the components of the study device (including lidocaine or any amide-based anesthetic), or history of allergies to any bovine collagen products, including but not limited to injectable collagen, collagen implants, hemostatic sponges, and collagen-based sutures.
* Undergone or planning to undergo desensitization injections to meat products.
* Unable to communicate or cooperate with the Investigator due to a language barrier (non-English speaking), poor mental development, or impaired cerebral function.
* Evidence of alcohol or drug abuse (Investigator opinion), or history of poor cooperation, non-compliance with medical treatment, or unreliability.
* Use of an investigation device, biologic or drug in the past 30 days, or is current participation in an experimental drug, biologic or device trial.
* A condition or situation that, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.
* Be an employee (or a relative of an employee) of the Investigator, Sponsor or representative of the Sponsor.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Male and Female
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Histopathology | 1 week
  Histopathologic examination of tissue samples to characterize PMMA induced collagen production in the dermis and deep dermis tissue.
Histopathology | 1 month
  Histopathologic examination of tissue samples to characterize PMMA induced collagen production in the dermis and deep dermis tissue.
Histopathology | 2 months
  Histopathologic examination of tissue samples to characterize PMMA induced collagen production in the dermis and deep dermis tissue.
Histopathology | 3 months
  Histopathologic examination of tissue samples to characterize PMMA induced collagen production in the dermis and deep dermis tissue.
Histopathology | 6 months
  Histopathologic examination of tissue samples to characterize PMMA induced collagen production in the dermis and deep dermis tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Seretta, Study Director — Suneva Medical
Locations (1):
- Call Suneva for Info, Danville, California, United States

IPD SHARING:
Plan to Share IPD: No